CLINICAL TRIAL: NCT05219617
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Carisbamate (YKP509) as Adjunctive Treatment for Seizures Associated With Lennox-Gastaut Syndrome in Children and Adults, With Optional Open-Label Extension
Brief Title: Investigate Efficacy and Safety of Carisbamate as Adjunctive Treatment for Seizures Associated With LGS in Children and Adults
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YKP509C003
Record Dates: First submitted 2022-01-06; First posted 2022-02-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Seizures; Lennox Gastaut Syndrome
Keywords: Seizures; Lennox Gastaut Syndrome; Pediatrics; Adults
MeSH Terms: conditions — Seizures; Lennox Gastaut Syndrome | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Intervention Model Description: This double-blind, randomized, placebo-controlled study will evaluate the efficacy of carisbamate 200 mg BID or the pediatric equivalent dose and 300 mg BID or the pediatric equivalent dose for the treatment of seizures associated with Lennox Gastaut syndrome in subjects 4 to 55 years of age.
Who Masked: Participant, Care Provider
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Carisbamate 200 mg BID arm (Experimental): Age: 4 to <12y* Titration: 2 mg/kg BID Maintenance: 4 mg/kg BID
  Age: ≥12 y Titration: 100 mg BID Maintenance: 200 mg BID
  Interventions: Drug: Carisbamate
- Carisbamate 300 mg BID arm (Experimental): Age: 4 to <12y* Titration: 2.75 mg/kg BID Maintenance: 5.5 mg/kg BID
  Age: ≥12 y Titration: 150 mg BID Maintenance: 300 mg BID
  Interventions: Drug: Carisbamate
- Placebo matched to 200 mg BID arm (Placebo Comparator): Age: 4 to <12y* Titration: Volume equivalent to 2 mg/kg BID Maintenance: Volume equivalent to 4 mg/kg BID
  Age: ≥12 y Titration: Volume equivalent to 100 mg BID Maintenance: Volume equivalent to 200 mg BID
  Interventions: Drug: Carisbamate
- Placebo matched to 300 mg BID arm (Placebo Comparator): Age: 4 to <12y* Titration: Volume equivalent to 2.75 mg/kg BID Maintenance: Volume equivalent to 5.5 mg/kg BID
  Age: ≥12 y Titration: Volume equivalent to 150 mg BID Maintenance: Volume equivalent to 300 mg BID
  Interventions: Drug: Carisbamate

INTERVENTIONS:
Drug: Carisbamate — Adolescent subjects 12 to 18 years old will receive the same dose as adults. Subjects 4 to < 12 years old in the carisbamate 200 mg BID arm will receive 4 mg/kg BID (not to exceed 200 mg BID [or a total of 400 mg per day]).
  Subjects 4 to < 12 years old in the carisbamate 300 mg BID arm will receive 5.5 mg/kg BID (not to exceed 300 mg BID [or a total of 600 mg per day]).

SUMMARY:
The primary objective is to evaluate the efficacy of carisbamate (YKP509) as adjunctive treatment in reducing the number of drop seizures (tonic, atonic, and tonic-clonic) compared with placebo in pediatric and adult subjects (age 4-55 years) diagnosed with Lennox Gastaut Syndrome (LGS).

DETAILED DESCRIPTION:
The secondary objectives are:

* To evaluate the efficacy of carisbamate (YKP509) as adjunctive treatment in reducing the total number of seizures compared with placebo in pediatric and adult subjects diagnosed with Lennox Gastaut Syndrome (LGS)
* Evaluate the safety, tolerability of carisbamate in the LGS population
* Evaluate steady-state pharmacokinetics of carisbamate in subjects with Lennox Gastaut.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a documented history of Lennox-Gastaut syndrome by:

   1. Evidence of more than one type of seizure, of which at least one should be an atonic or tonic seizure
   2. History of an electroencephalogram (EEG) reporting diagnostic criteria for LGS (abnormal background activity accompanied by slow, spike and wave pattern <3.0 Hz)
   3. History of developmental delay
2. Male or female subjects
3. Subjects must be age 4-55 years at the time of consent/assent
4. Must have been <11 years old at the onset of LGS
5. Subjects must have experienced at least 2 drop seizures with potential to fall (tonic, atonic, tonic-clonic) during the 4-week Baseline period preceding randomization (minimum of 4 drop seizures in the first two weeks and 4 in the last two weeks). Drop seizures are defined as a seizure involving the entire body, trunk, or head that led or could have led to a fall, injury, slumping in a chair, or hitting the subject's head on a surface. All drop seizure types must be countable (either as isolated seizures or as countable isolated seizures in a cluster).
6. Subjects must have been receiving 1 to 4 concomitant anti-seizure medications (ASMs) at a stable dose for at least 4 weeks before Visit 1
7. If not taking Epidiolex, subjects may take other approved cannabidiol or over the counter cannabidiol products. If taking cannabidiol other than Epidiolex, consult Medical Monitor to determine if it counts as a concomitant ASM.
8. Dietary therapy and any CNS stimulator settings must be stable for 4 weeks prior to baseline and maintain stable regimen throughout the study. The dietary therapy and CNS stimulators are not counted as an ASM.
9. Parents or caregivers must be able to keep accurate seizure diaries
10. Subject is either not of childbearing potential, defined as premenarchal, postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), if of childbearing potential, must comply with an acceptable method of birth control during the study, for at least 4 weeks prior to study entry and for 4 weeks following completion of the study, if able.
11. Subject and/or caregiver(s)/legal representative must be willing and able to give informed assent/consent for participation in the study
12. Subject and their caregiver must be willing and able (in the investigator's opinion) to comply with all study requirements
13. History of COVID-19 vaccination is permitted

Exclusion Criteria:

1. Etiology of subject's seizures is a progressive neurologic disease. Subjects with tuberous sclerosis will not be excluded from study participation, unless there is a progressive brain tumor
2. Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal disease, hepatic disease) that in the opinion of the investigator(s) could affect the subject's safety or study conduct
3. Subjects who were on adrenocorticotropic hormone (ACTH) therapy in the 6 months prior to baseline
4. Subject on dietary therapy for less than 4 weeks prior to screening visit (Visit 1) or suffers from frequent stooling
5. Current use of felbamate with less than 18 months of continuous exposure
6. Concomitant use of vigabatrin: subjects who took vigabatrin in the past must be discontinued for at least 5 months before Visit 1 and must have documentation showing no evidence of a vigabatrin-associated clinically significant abnormality in an automated visual perimetry test, if able.
7. Subject who had a history of hypoxia which needed emergency resuscitation within 12 months prior to baseline
8. Status epilepticus within 12 weeks prior to Visit 1
9. Any clinically significant illness (including COVID-19) in the 4 weeks prior to Visit 1, as evaluated by the Investigator
10. Subject has clinically significant abnormal laboratory values, in the investigator's opinion, at Visit 1 or time of randomization (Visit 2)
11. Subject has a history of any serious drug-induced hypersensitivity, e.g., toxic epidermal necrolysis, or Drug Reaction with Eosinophilia and Systemic Symptoms [DRESS]) or any drug-related rash requiring hospitalization
12. Vagus Nerve Stimulation (VNS), Deep Brain Stimulation (DBS), Responsive Neurostimulator System (RNS) or other neurostimulation for epilepsy device implanted or activated <5 months year prior to enrollment. Stimulation parameters that have been stable for <4 weeks, or Battery life of unit not anticipated to extend for duration of trial.
13. Subject is pregnant, may be pregnant, lactating or planning to be pregnant
14. Any suicidal ideation with intent, with or without a plan within 6 months before Visit 2 (i.e., answering "Yes" to questions 4 or 5 in the Suicidal Ideation section of the age- specific Columbia-Suicide Severity Rating Scale (C-SSRS) in subjects aged 6 and above who are able to be evaluated
15. Any suicidal behavior within 2 years before Visit 2 (i.e., answering YES to any question in the Suicidal behavior section of the age-specific Columbia-Suicide Severity Rating Scale (C-SSRS) in subjects aged 6 and above who are able to be evaluated.
16. Evidence of significant active hepatic disease. Stable elevations of liver enzymes (alanine aminotransferase (ALT), and aspartate aminotransferase (AST)) due to concomitant medication(s) will be allowed if they are <3 x ULN
17. Subject with total bilirubin [TBL] >2 x ULN (except for Gilbert's syndrome).
18. Active viral hepatitis (B or C) as demonstrated by positive serology at the Screening visit (Visit 1)
19. History of positive antibody/antigen test for human immunodeficiency virus (HIV)
20. If taking Epidiolex, subject may not use other approved cannabidiol or over the counter cannabidiol products
21. Scheduled for epilepsy-related surgery, VNS insertion, or any other stimulators/surgery during the projected course of the study
22. Subject who has taken or used any investigational drug or device in the 4 weeks prior to the screening visit (Visit 1)
23. Concomitant use of medications known to be strong inducers of cytochrome P450 (CYP3A) including, but not limited to: phenobarbital, phenytoin, carbamazepine, primidone, rifampin, troglitazone, St. John's Wort, efavirenz, nevirapine, glucocorticoids (other than topical usage), modafinil, pioglitazone, and rifabutin
24. Evidence of cardiac disease, including unstable angina, myocardial infarction, within the past 2 years, uncontrolled heart failure, major arrhythmias, congenital short QT syndrome
25. Subject with a short QTc interval (<340 msec) or long QTc interval (>460 msec) as confirmed by a repeated electrocardiogram (ECG)
26. Benzodiazepine rescue administered on average more than once a week in the month before Visit 1
27. Previous exposure to carisbamate or sensitivity/allergy to components of the oral suspension.

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome will be the percentage change from baseline in the total frequency (average per 28 days) of countable drop seizures with potential to fall (tonic, atonic, tonic-clonic) seizures during the double-blind treatment period. | 3 years
  Efficacy of Carisbamate YKP509

SECONDARY OUTCOMES:
The percentage of subjects with at least a 50% reduction from baseline in the total frequency of drop seizures (tonic, atonic, tonic-clonic) during the double-blind treatment period. | 3 years
  Efficacy of Carisbamate YKP509
Percentage change from baseline in the frequency of all types of seizures (total seizures) during the double-blind treatment period. | 3 years
  Efficacy of Carisbamate YKP509
Subject/Caregiver Global Impression of Change (S/CGIC) in overall condition score at the last visit. | 3 years
  Efficacy of Carisbamate YKP509- Scoring will be from 1 to 7 with 1 (very much improved) to 7 (very much worse)

OTHER OUTCOMES:
Percentage change from baseline in the 28-day frequency of: drop seizures (tonic, atonic, tonic-clonic); non-drop seizures (myoclonic seizures, atypical absence); total seizures during the maintenance phase of the double-blind treatment period. | 3 years
  Efficacy of Carisbamate YKP509
Percentage change from baseline in non-drop seizures (myoclonic seizures, atypical absence) frequency per 28 days during the during the double-blind treatment period. | 3 years
  Efficacy of Carisbamate YKP509
The percentage of subjects with at least a 50% reduction from baseline in the total frequency of drop seizures (tonic, atonic, tonic-clonic) during the maintenance phase of the double-blind treatment period. | 3 years
  Efficacy of Carisbamate YKP509
Proportion of subjects with a 75%, 90% and 100% response rate for drop seizures (tonic, atonic, tonic-clonic), non-drop seizures, and total seizures during the double-blind treatment period. | 3 years
  Efficacy of Carisbamate YKP509
Proportion of subjects with a 75%, 90% and 100% response rate for drop seizures (tonic, atonic, tonic-clonic), non-drop seizures, and total seizures during the maintenance phase of the double-blind treatment period. | 3 years
  Efficacy of Carisbamate YKP509

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kamin, MD, Study Director — SK Life Science, Inc.
Locations (71):
- United States (22):
  - Stanford University Hospital, Palo Alto, California
  - University of Florida Health Science Center, Jacksonville, Florida
  - AdventHealth, Orlando, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Axcess Medical Research, Wellington, Florida
  - Consultants in Epilepsy and Neurology PLLC, Boise, Idaho
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri School of Medicine, Columbia, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - St. Peters Hospital, New Brunswick, New Jersey
  - Montefiore, The Bronx, New York
  - Duke University Clinical Research at Pickett Road, Durham, North Carolina
  - Wake Forest University - School of Medicine, Winston-Salem, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Austin Epilepsy Care Center - Clinic/Outpatient Facility, Austin, Texas
  - Neurology Consultants of Dallas, PA - Hospital, Dallas, Texas
  - Virginia Epilepsy and Neurodevelopmental Clinic at WNC, Winchester, Virginia
- Argentina (2):
  - Hospital de Ninos de La Santisma Trinidad, Córdoba, Córdoba Province
  - Resolution Psychopharmacology Research Institute, Mendoza, Mendoza Province
- Australia (4):
  - Austin Hosptial, Heidelberg
  - Alfred Health, Melbourne
  - Perth's Children Hospital, Nedlands
  - Queensland Children's Hospital, South Brisbane
- Colombia (5):
  - Fundacion Hospital Universidad del Norte, Barranquilla
  - Fundacion Valle del Lili/Clinic - Outpatient, Cali
  - CliniSalud del Sur S.A.S - Centro de Investigación, Envigado
  - Hospital Pabloe Tubon Uribe, Medellín
  - Institutio Neurologico de Colombia, Medellín
- Germany (2):
  - Universitatsklinikum Erangen, Erlangen, Bavaria
  - Kleinwachau Sächsisches Epilepsiezentrum, Radeberg, Saxony
- Iaso Children's Hospital, Marousi, Attica, Greece
- Hungary (2):
  - Orszagos Mentalis, Ideggyogyaszati es Idegsebezeti Intezet, Budapest
  - Semmelweis Egyetem Idegsebeszeti es Neurointervencios Klinika, Budapest
- Israel (4):
  - Tela Viv Sourlasky Medical Center, Tel Aviv, Tel Aviv
  - Soroka University Medical Centre, Beersheba
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (6):
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genoa, Liguria
  - ASST Fatebenefratelli Sacco - Ospedale dei Bambini Vittore Buzzi, Milan, Lombardy
  - Fondazione IRCCS Di Rilievo Nazionale Instituto, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Verona
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence
  - ASST Santi Paolo E Carlo - Azienda Universitaria-Polo Universitaria - San Paolo, Milan
- Mexico (3):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Neurociencias Estudios Clinicos S.C., Culiacán
  - Clinstile, S.A. de C.V., Mexico City
- Poland (2):
  - Szpital Kliniczny im.H.Swiecickiego Uniwersytetu Medycznego im.K.Marcinkowskiego w Poznaniu-Dluga1/2, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Plejady, Krakow
- Portugal (4):
  - Centro Hospitalar de Lisboa Norte, EPE, Lisbon, Lisbon District
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Sao Francisco Xavier, Lisbon, Lisbon District
  - Centro Hospitalar de Sao Joao, EPE, Porto, Porto District
  - Hospital Garcia de Orta, Almada, Setúbal District
- Serbia (5):
  - Childrens University Hospital, Belgrade, Belgrade
  - University Clinical Center of Serbia - PPDS, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
  - Children and Youth Health Care Institute of Vojvodina, Novi Sad
- South Korea (3):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (3):
  - Hospital Sant Joan de Deu - PIN, Esplugues de Llobregat, Barcelona
  - Hospital Infantil Universitario Niño Jesus - PIN, Madrid
  - Hospital Ruber Internacional (Grupo Quironsalud), Madrid
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided